CLINICAL TRIAL: NCT02669992
Title: Loop Ileostomy Closure.Stapled or Hand-sewn Anastomoses? Suture or Mesh Closure of the Stoma Site in the Abdominal Wall. A Prospective Randomised Multicenter Trial.
Brief Title: Loop Ileostomy Closure:Stapled or Hand-sewn Anastomoses? Suture or Mesh Closure of the Stoma Site?
Acronym: LISTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Ulrik Lindforss, Associate professor, Karolinska University Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2015/321-31/1
Record Dates: First submitted 2015-12-08; First posted 2016-02-01 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Rectal Neoplasm
Keywords: Ileostomy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Stapled anastomosis (Experimental): Stapled anastomosis by the use of commercially available linear stapler device
  Interventions: Procedure: Stapled or Hand-sewn anastomosis
- Hand-sewn anastomosis (Active Comparator): Hand-sewn by the use of a resorbable monofilament suture
  Interventions: Procedure: Stapled or Hand-sewn anastomosis
- Abdominal wall mesh closure (Experimental): Closure by the use of a mesh low-weight net device
  Interventions: Procedure: Mesh or suture stoma site closure
- Abdominal wall suture closure (Active Comparator): Closure by the use of slowly absorbing monofilament suture
  Interventions: Procedure: Mesh or suture stoma site closure

INTERVENTIONS:
Procedure: Stapled or Hand-sewn anastomosis — Randomization between stapled or hand-sewn anastomosis
  Arms: Hand-sewn anastomosis; Stapled anastomosis
Procedure: Mesh or suture stoma site closure — Randomization between suture or Mesh closure of the stoma site
  Arms: Abdominal wall mesh closure; Abdominal wall suture closure

SUMMARY:
There are severel problems associated with the closing of a temporary loop-ileostomy after surgery for rectal cancer. The purpose of this study is to answer two questions:

1. The choice of anastomotic method - does it influence the postoperative course?
2. The use of a prophylactic mesh when closing the stoma site - will there be less hernias?

DETAILED DESCRIPTION:
Postoperative complications after closure of a temporary loop ileostomy after rectal cancer surgery are common. In this study the investigators propose the hypothesis that a stapled anastomotic technique will decrease postoperative small bowel obstruction and a mesh closure of the stoma site in the abdominal wall will decrease hernia formation.

All patients will be randomized to stapled or hand-sewn anastomosis. The randomization to mesh or suture closure of the abdominal wall is optional.

The stapled anastomotic technique is performed by the use of a linear staple device and the hand-sewn technique with a running seromuscular monofilament suture.

The stoma site has two options and will be closed either by the use of mesh (lightweight), positioned under the muscle (retromuscular), or just by long-lasting suture. The anterior fascia of the rectus as well as the skin are closed by the use of running monofilament longlasting sutures, the latter in a pursestring procedure.

ELIGIBILITY:
Inclusion Criteria:

* loop ileostomy after rectal cancer surgery
* loop ileostomy closure is permitted and possible according to clinical practice

Exclusion Criteria:

* patient unable to understand written or oral information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with postoperative bowel obstruction | 30 days
  Postoperative bowel obstruction within 30 Days, detected clinically or by the use of x-ray
Number of participants with postoperative stoma site hernia | 2 year
  Herni postoperatively on the site of previous stoma detected within 2 years

SECONDARY OUTCOMES:
Number of participants with postoperative complications | 30 days
Postoperative Hospital stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Lindforss, A.P, Principal Investigator — Karolinska University Hospital
Locations (11):
- Sweden (11):
  - Sahlgrenska Universitetssjukhuset, Östra sjukhuset, Gothenburg
  - Centralsjukhuset Karlstad, Karlstad
  - Sunderby Sjukhus, Luleå
  - Lycksele lasarett, Lycksele
  - Norrtälje sjukhus, Norrtälje
  - Östersunds sjukhus, Östersund
  - Skellefteå lasarett, Skellefteå
  - Danderyds sjukhus, Stockholm
  - Karolinska universitetssjukhuset, Stockholm
  - Norrlands Universitets Sjukhus, Umeå
  - Region Gotland, Visby

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gustavsson K, Gunnarsson U, Jestin P. Postoperative complications after closure of a diverting ileostoma--differences according to closure technique. Int J Colorectal Dis. 2012 Jan;27(1):55-8. doi: 10.1007/s00384-011-1287-4. Epub 2011 Aug 16. PMID 21845418
- [Background] Gong J, Guo Z, Li Y, Gu L, Zhu W, Li J, Li N. Stapled vs hand suture closure of loop ileostomy: a meta-analysis. Colorectal Dis. 2013;15(10):e561-8. doi: 10.1111/codi.12388. PMID 24033921
- [Background] Rubio-Perez I, Leon M, Pastor D, Diaz Dominguez J, Cantero R. Increased postoperative complications after protective ileostomy closure delay: An institutional study. World J Gastrointest Surg. 2014 Sep 27;6(9):169-74. doi: 10.4240/wjgs.v6.i9.169. PMID 25276286
- [Background] Akiyoshi T, Fujimoto Y, Konishi T, Kuroyanagi H, Ueno M, Oya M, Yamaguchi T. Complications of loop ileostomy closure in patients with rectal tumor. World J Surg. 2010 Aug;34(8):1937-42. doi: 10.1007/s00268-010-0547-8. PMID 20372898
- [Background] Chude GG, Rayate NV, Patris V, Koshariya M, Jagad R, Kawamoto J, Lygidakis NJ. Defunctioning loop ileostomy with low anterior resection for distal rectal cancer: should we make an ileostomy as a routine procedure? A prospective randomized study. Hepatogastroenterology. 2008 Sep-Oct;55(86-87):1562-7. PMID 19102343
- [Background] Loffler T, Rossion I, Bruckner T, Diener MK, Koch M, von Frankenberg M, Pochhammer J, Thomusch O, Kijak T, Simon T, Mihaljevic AL, Kruger M, Stein E, Prechtl G, Hodina R, Michal W, Strunk R, Henkel K, Bunse J, Jaschke G, Politt D, Heistermann HP, Fusser M, Lange C, Stamm A, Vosschulte A, Holzer R, Partecke LI, Burdzik E, Hug HM, Luntz SP, Kieser M, Buchler MW, Weitz J; HASTA Trial Group. HAnd Suture Versus STApling for Closure of Loop Ileostomy (HASTA Trial): results of a multicenter randomized trial (DRKS00000040). Ann Surg. 2012 Nov;256(5):828-35; discussion 835-6. doi: 10.1097/SLA.0b013e318272df97. PMID 23095628